CLINICAL TRIAL: NCT00202774
Title: Phase III, Multicenter, Ramdomised, Open-label, Study to Evaluate the Safety and Efficacy of Combination Therapy With XELOX vs. Oxaliplatin and 5-FU CI as First Line Treatment in Advanced or Metastatic Colorectal Cancer
Brief Title: Safety and Efficacy Study of XELOX vs. Oxaliplatin+5-FU CI as First Line Treatment in Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Spanish Cooperative Group for the Treatment of Digestive Tumours (TTD) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-TTD-01
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2023-04-12 (Actual); Status verified 2019-04

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer, capecitabine, oxaliplatin, 5-fluorouracil
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Oxaliplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: (capecitabine, oxaliplatin, 5-fluorouracil)

SUMMARY:
The purpose of this study is to determine time to disease progression of combination therapy with capecitabine and oxaliplatin (XELOX) vs. oxaliplatin and 5-fluorouracil in continous infusion (5-FU CI) as first line treatment in advanced or metastatic colorectal cancer

DETAILED DESCRIPTION:
The purpose of this study is to determine time to disease progression of combination therapy with capecitabine and oxaliplatin (XELOX) vs. oxaliplatin and 5-fluorouracil in continous infusion (5-FU CI) as first line treatment in advanced or metastatic colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

Written informed consent. Men and women > or = 18 years Karnofsky functional status >or=70% at the time of enrollment in study Histologically confirmed diagnosis of CRC Patients must not have received chemotherapy (exception: adjuvant treatment > 12 months following conclusion of treatment) Presence of at least one lesion detectable by two-dimensional measurement.. Life expectancy greater than 3 months.

Exclusion Criteria:

Pregnant or nursing woman Prior administration of systemic immunotherapy, chemotherapy (exception: 5-FU as adjuvant treatment > 12 months following conclusion of treatment) Evidence of allergic reaction to any of the treatment components Clinically relevant myocardial disease or history of myocardial infarction in the past 12 months Documented or suspected cerebral and/or leptomeningeal metastases. Prior malignant tumour in past 5 years, except history of basal cell skin carcinoma or pre-invasive cervical carcinoma.

Neutrophil count < 1.5 x 109/l , platelets < 100 X 109/l serum creatinine > 1.5 x ULN. Total bilirubin count > 2 x ULN Alkaline Phosphatase > > 2.5 x ULN (> 5 x ULN if there are hepatic metastases) Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) > 2.5 x ULN (> 5 x ULN if there are hepatic metastases, > 10 x ULN if there are bone metastases) Creatinine clearance < 30 ml/min Surgery within 4 weeks prior to enrollment in the study. Any investigational drug during the 4 weeks prior to enrolment. Uncontrolled active infection Any medical or psychological disorder which, in the opinion of the investigator, does not allow the patient to conclude the study or sign the informed consent

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2002-04; Primary Completion 2004-08 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Determine time to disease progression

SECONDARY OUTCOMES:
Determine safety of combination, objetive response rate, time to onset of response , duration of response, time to treatment failure, one year survival time, overall survival time

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Aranda, Study Chair — Spanish Cooperative Group for Gastrointestinal Tumour Therapy (TTD); Eduardo Díaz-Rubio, Study Chair — Spanish Cooperative Group for Gastrointestinal Tumour Therapy (TTD)
Locations (1):
- Spanish Cooperative Group for Gastrointestinal Tumour Therapy (TTD), Madrid, Spain